CLINICAL TRIAL: NCT05215821
Title: HOMA Estimated Insulin Resistance as a Marker for Angiographic Severity of Coronary Artery Disease in Non Diabetic & Non Obese Patients.
Brief Title: Insulin Resistance and Severity of Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ahmed Altaher, clinical professor, Sohag University
Other Study IDs: Soh-Med-22-01-42
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group1: subjects with evidence of insulin resistance estimated by high HOMA level
- group 2: subjects without insulin resistance estimated by normal HOMA level

SUMMARY:
this is an observertional study aimed at Study the association between Insulin resistance estimated by HOMA and Angiographic Severity of Coronary Artery Disease in Non Diabetic & Non Obese Patients.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing coronary angiography (CA) for ACS or stable angina in the Catheterization Laboratory of internal Medicine department and El Noor specialized cardiac center at the study period.

Exclusion Criteria:

* age < 18 years,
* pregnancy or breastfeeding,
* BMI >30 Kg/m2 and
* presence of pre-diabetes or overt diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing coronary angiography due to suspected coronary artery disease
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
HOMA IR level estimated by Two-site immunoenzymometric assay | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali mo Altaher, lecturer, Principal Investigator — Sohag faculty of medicine
Locations (1):
- Sohag uniersity hosoital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided